CLINICAL TRIAL: NCT05888376
Title: A Post-Market Clinical Performance and Safety Evaluation of GamCath HighFlow Dolphin Protect Catheter
Status: Completed | Type: Observational
Sponsor: Vantive Health LLC (Industry)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: BXU565389
Record Dates: First submitted 2023-05-15; First posted 2023-06-05 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: AKI - Acute Kidney Injury; Acute Renal Failure; CKD; ESRD
Keywords: extracorporeal blood purification; continuous renal replacement therapy
MeSH Terms: conditions — Acute Kidney Injury; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Consecutive CKD including ESRD treatments: Consecutive retrospective treatments across all sites with a diagnosis of CKD, including ESRD
  Interventions: Device: Vascular access catheter to support dialysis or CRRT
- Consecutive treatments with minimum hospital stay of 20 days: Consecutive retrospective treatments across all sites with a minimum hospital stay of days (excluding cases previously identified; may be acute or chronic disease)
  Interventions: Device: Vascular access catheter to support dialysis or CRRT
- Consecutive acute/chronic kidney disease treatments: Consecutive retrospective treatments across all sites with acute or chronic disease (excluding cases previously identified)
  Interventions: Device: Vascular access catheter to support dialysis or CRRT

INTERVENTIONS:
Device: Vascular access catheter to support dialysis or CRRT — A specialised vascular access catheter to support bi-directional blood flow at high rates to allow extracorporeal removal of toxins by dialysis or CRRT

SUMMARY:
The goal of this retrospective chart review is to obtain clinical safety and performance data for the GamCath HighFlow Dolphin Protect Catheter in patients with acute kidney injury, acute renal failure, or chronic kidney disease.

The main questions to answer are:

1. Duration of catheter use (survival)
2. Reason(s) for catheter removal

DETAILED DESCRIPTION:
The objective of this retrospective chart review is to obtain clinical safety and performance data for the GamCath HighFlow Dolphin Protect Catheter related to the duration of use (catheter survival) throughout its lifetime.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age at the time of catheter insertion.
* Patients diagnosed with AKI, ARF, and/or CKD (including end-stage renal disease [ESRD]).
* Patients who required vascular access to perform extracorporeal blood purification using GamCath HighFlow Dolphin Protect Catheter inserted by a physician in the subclavian, jugular, or femoral veins.

Exclusion Criteria:

* Patients who required the GamCath HighFlow Dolphin Protect Catheter for any indication other than extracorporeal blood purification.
* Patients who had a local infection at the vascular access site prior to catheter insertion.
* Patients who required surgical intervention (e.g., cutdown procedure) for GamCath HighFlow Dolphin Protect Catheter placement.
* Patients who had a prior catheter in place at the same vascular access site (i.e., R/L jugular vein, R/L femoral vein, R/L subclavian vein) within the last 7 days.
* Patients who do not have complete patient records to support the primary endpoint analyses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be collected from records of adult patients in whom the GamCath HighFlow Dolphin Protect Catheter was inserted as a vascular access to perform extracorporeal blood purification from 2018 to most recent.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Catheter Survival | From date of catheter insertion until the date of catheter removal or patient transfer or discharge or death, whichever occurs first, assessed up to 12 weeks
  Confirm catheter lifetime related to GamCath HighFlow Dolphin Protect Catheter duration of use to support PMCF ongoing performance data
Reason(s) for Catheter Removal | Within 72 hours of catheter removal or patient transfer or discharge or death, whichever occurs first, assessed up to 12 weeks
  Collect additional real-world use data describing the reason(s) for GamCath HighFlow Dolphin Protect Catheter removal to support PMCF ongoing product safety performance

SECONDARY OUTCOMES:
Adverse Events | From date of catheter insertion until the date of catheter removal or patient transfer or discharge or death, whichever occurs first, assessed up to 12 weeks
  Collect real-world use data describing adverse events potentially related to the study catheter or catheter insertion/removal procedures

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Dąbrowski, Prof MD PhD, Principal Investigator — Independent Public Clinical Hospital No. 4, Lublin; Marek Winiarz, MD, Principal Investigator — Independent Public Health Care Unit, Łęczna
Locations (2):
- Poland (2):
  - Independent Public Hospital No. 4, Lublin, Lublin
  - Independent Public Health Care Unit, Łęczna, Łęczna

IPD SHARING:
Plan to Share IPD: No
The Sponsor is committed to sharing clinical trial data with external medical experts and scientific researchers in the interest of advancing public health. As such, the Sponsor will supply anonymized Individual Patient Datasets (IPD) and supporting documents (synopsis of clinical study reports, protocol and SAP). Research requests will be reviewed by qualified medical and scientific experts within the company. If the Sponsor agrees to the release of clinical data for research purposes, the requestor will be required to sign a data sharing agreement (DSA) in order to ensure protection of patient confidentiality and any intellectual property rights of the Sponsor prior to the release of any data.